CLINICAL TRIAL: NCT05372601
Title: The Effect of Galacto-oligosaccharides (GOS) on Self-perceived Stress in Apparently Healthy But Stressed Dutch Women: Randomized Controlled Study
Brief Title: Prebiotics and Stress Reduction in Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: FrieslandCampina (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Stress Defense
Record Dates: First submitted 2022-02-11; First posted 2022-05-13 (Actual); Last update posted 2024-03-04 (Actual); Status verified 2024-03

CONDITIONS: Stress, Psychological
MeSH Terms: conditions — Stress, Psychological | interventions — maltodextrin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Relax+ (Experimental): Relax+ consists of a powder containing a blend of two prebiotics.
  Interventions: Dietary Supplement: Relax+
- Placebo (Placebo Comparator): The placebo contains maltodextrin.
  Interventions: Dietary Supplement: Maltodextrin

INTERVENTIONS:
Dietary Supplement: Relax+ — Prebiotics, daily administered
  Arms: Relax+
Dietary Supplement: Maltodextrin — Placebo, daily administered
  Arms: Placebo

SUMMARY:
In modern life, many people state to experience stress. Women compared to men report more and higher levels of stress. Recent research found that supplementation of galactose-oligosaccharides (GOS) resulted in reduced anxiety levels in British female students with higher anxiety scores at baseline in self-reported trait anxiety. Moreover, supplementation of probiotics in germ-free rodents resulted in reduced levels of circulating corticosterone (cortisol in humans). These findings illustrate the potential of prebiotic supplementation, through the microbiota-gut-brain (MGB) axis, to improve mental health and wellbeing.

The present study aims to study the effect of oligosaccharides on self-perceived stress.

ELIGIBILITY:
Inclusion Criteria:

* Apparently healthy women
* Moderate or high stress level; DASS42 stress sub-score ≥19
* Age between 25 and 45 years
* Body mass index (BMI) between 18.5 and 30 kg/m2
* Access to internet and a smart phone

Exclusion Criteria:

* Any metabolic, gastrointestinal, inflammatory or chronic disease
* History of gastro-intestinal surgery or having (serious) gastrointestinal discomfort
* Use of supplement to relief stress during or within 2 weeks prior to the start of the study
* Use of pre- and/or probiotics during the study (except for the study product) or within 4 weeks prior to the start of the study
* Use of medication that may influence the study results, such as laxatives
* Self-reported and/or clinical lactose intolerance
* Self-reported and/or active cow's milk protein allergy
* Pregnant or lactating (or having the wish to become pregnant during the study period, self-reported)
* Having used antibiotics in the 6 months prior to the start of the study

Ages: 25 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 124 (Actual)
Dates: Start 2022-02-17 (Actual); Primary Completion 2022-06-18 (Actual); Study Completion 2022-06-18 (Actual)

PRIMARY OUTCOMES:
Perceived stress | 28 days
  The difference in absolute stress sub-score after the product intervention between the product groups (using the Depression Anxiety Stress Scale (DASS-42)), in which a lower score corresponds with a lower stress level

CONTACTS AND LOCATIONS:
Overall Officials: Reina S Tjoelker, MSc, Principal Investigator — FrieslandCampina
Locations (1):
- FrieslandCampina Research and Development, Wageningen, Netherlands

IPD SHARING:
Plan to Share IPD: No